CLINICAL TRIAL: NCT02984644
Title: Paradoxical Stimulation of Hepatic Glucose Production With Dapagliflozin (P2)
Brief Title: Paradoxical Stimulation of Hepatic Glucose Production With Dapagliflozin
Acronym: AZ11040
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20160586H
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Type II; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): 32 subjects will receive dapagliflozin 10mg
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): 16 subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Three 5-hour measurements (after dapagliflozin 10mg administration) of endogenous glucose production (EGP) will be performed on separate days.
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Three 5-hour measurements (after placebo administration) of endogenous glucose production (EGP) will be performed on separate days.
  Other Names: Placebo for Dapagliflozin
  Arms: Placebo

SUMMARY:
To determine the role of plasma glucagon and insulin in the rise of endogenous glucose production (EGP) following the SGLT2 inhibition.

DETAILED DESCRIPTION:
The increase in plasma glucagon conc and/or decrease in plasma insulin conc in response to glucosuria is (are) important signal(s) responsible, at least in part, for the increase in EGP, which the investigators anticipate will be derived primarily from the liver. Insulin and glucagon are powerful regulators of HGP. Therefore, the investigators anticipate that, at least in part, an increase in HGP secondary to the rise in plasma glucagon concentration and decrease in plasma insulin concentration in response to dapagliflozin-induced glucosuria will account for the majority of increase in EGP in both NGT and T2DM subjects. This study will define whether the increase in plasma glucagon and/or the decrease in plasma insulin are the trigger to stimulate EGP. Eligible subjects will receive three 5-hour measurements of endogenous glucose production (EGP), which is the biosynthesis of new glucose, with administration of study drug after a 3-hour tracer equilibration period. Hepatic glucose production (HGP), which is the net release of glucose from the liver, will be measured for 5 hours after drug administration to allow sufficient time for a significant increase in HGP above baseline after dapagliflozin administration (10). In study 1, HGP will be measured for 5 hours after dapagliflozin (10 mg) or placebo administration. This is the control study. The investigators expect to observe the "paradoxical" rise in EGP following dapagliflozin. Study 2 will be performed under glucose clamp conditions (i.e. maintaining the plasma glucose concentration stable at each subject's fasting level). This study will define whether the decline in plasma glucose concentration is the trigger to stimulate EGP. Study 3 will be performed under pancreatic clamp conditions (maintaining the plasma glucagon and insulin concentrations constant at the basal level). This study will define whether the increase in plasma glucagon and/or the decrease in plasma insulin are the trigger to stimulate EGP. Subjects will be randomized in a 2:1 ratio; 32 subjects will receive dapagliflozin and 16 subjects will receive placebo. Each study will be performed on a separate day, after a 10-12 hour overnight fast within 1-2 week period. Following studies 1-3, subjects will return for a renal (kidney) MRI-measurement to record kidney size.

ELIGIBILITY:
Inclusion Criteria:

* T2DM according to ADA criteria-HbA1C < 8.0%
* BMI = 25-35 kg/m2
* Subjects must be in good general health as determined by physical exam, medical history, blood chemistries, CBC, TSH, T4, EKG and urinanalysis
* Body weight has been stable (± 3 lbs) over the preceding three months
* Do not participate in an excessively heavy exercise program
* Taking stable dose (more than 3 months) of monotherapy or combination therapy with metformin and/or a sulfonylurea

Exclusion Criteria:

* Subjects taking drugs known to affect glucose metabolism (other than metformin and sulfonylurea) will be excluded
* Individuals with evidence of proliferative diabetic retinopathy, plasma creatinine >1.4 females or >1.5 males, or 24-hour urine albumin excretion > 300 mg will be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD,PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg
  Dapagliflozin: Three 5-hour measurements (after dapagliflozin 10mg administration) of endogenous glucose production (EGP) will be performed on separate days.
- Placebo: Subjects will receive placebo
  Placebo: Three 5-hour measurements (after placebo administration) of endogenous glucose production (EGP) will be performed on separate days.
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (2) | 53 (2) | 54 (2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 30 participants were randomized: 20 to the Dapagliflozin and 10 to the placebo arm of the study
  Participants
    Female | 8 | 3 | 11
    Male | 12 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 18
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 12 | 4 | 16
  Caucasian | 7 | 2 | 9
  African American | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Change in Plasma Glucose (mg/dL): Study 1
Description: Change from baseline to the last hour of the study (240-300 minutes) in plasma glucose concentration
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Dapagliflozin 10mg: Change in plasma glucose concentration to show effect of Dapagliflozin on EGP (endogenous glucose production)
- Placebo: Change in plasma glucose concentration after placebo administration
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 20 | 10
mg/dl | -29 (4) | -17 (3)

2. Primary Outcome: Change in Plasma Glucose Measurement Using a Glucose Clamp: Study 2
Description: Change from baseline to the last hour of the study (240-300 minutes) in plasma glucose for study 2: EGP plus glucose clamp. The glucose clamp technique is achieved by increase plasma glucose concentration to 125 mg/dl above basal levels by a continuous infusion of glucose. This hyperglycemic plateau is maintained by adjustment of a variable glucose infusion, based on the rate of insulin secretion and glucose metabolism. Because the plasma glucose concentration is held constant, the glucose infusion rate is an index of insulin secretion and glucose metabolism. The 3-3H-glucose infusion will be started at 6 AM to measure the basal rate of EGP. After a 3 hour tracer equilibration period (at 9 AM) subjects will receive dapagliflozin (10 mg) or placebo, and the plasma glucose conc will be measured every 5 minutes for 5 hours (from 9AM to 2 PM)
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Dapagliflozin 10mg: Change in plasma glucose concentration to show effect of Dapagliflozin on EGP (endogenous glucose production) using a glucose clamp
- Placebo: Change in plasma glucose concentration after placebo administration using a glucose clamp
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 20 | 10
mg/dl | 3 (1) | 1 (1)

3. Primary Outcome: Change in Plasma Glucose Using a Pancreatic Clamp: Study 3
Description: Change from Baseline to the last hour of the study (240-300 minutes) in plasma glucose using a pancreatic clamp. In this study, EGP will be measured as described in Study 1 and plasma insulin and glucagon concentrations will be clamped at the basal level using the pancreatic clamp technique. Plasma glucose concentration will be allowed to decrease spontaneously after dapagliflozin or placebo administration. Somastatin will be infused with glucagon and insulin to replace basal plasma glucagon and insulin until study end.
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Dapagliflozin 10mg: Change in plasma glucose concentration to show effect of Dapagliflozin on plasma glucose concentration
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 20 | 10
mg/dl | -30 (4) | -7 (5)

4. Primary Outcome: Change in EGP: Study 1
Description: Change from baseline to the last hour of the study (240-300 minutes) in EGP
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/kg.min
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
mg/kg.min | 0.10 (0.1) | -0.56 (0.11)

5. Primary Outcome: Change in EGP With Glucose Clamp: Study 2
Description: Change from baseline to the last hour of the study (240-300 minutes) in EGP using a glucose clamp. The glucose clamp technique is achieved by increase plasma glucose concentration to 125 mg/dl above basal levels by a continuous infusion of glucose. This hyperglycemic plateau is maintained by adjustment of a variable glucose infusion, based on the rate of insulin secretion and glucose metabolism. Because the plasma glucose concentration is held constant, the glucose infusion rate is an index of insulin secretion and glucose metabolism. The 3-3H-glucose infusion will be started at 6 AM to measure the basal rate of EGP. After a 3 hour tracer equilibration period (at 9 AM) subjects will receive dapagliflozin (10 mg) or placebo, and the plasma glucose conc will be measured every 5 minutes for 5 hours (from 9AM to 2 PM)
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/kg.min
Groups:
- Dapagliflozin 10mg: Change in EGP (endogenous glucose production) after dapagliflozin administration
- Placebo: Change in EGP concentration after placebo administration
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 20 | 10
mg/kg.min | -0.57 (0.12) | -1.28 (0.172)

6. Primary Outcome: Change in EGP With Pancreatic Clamp: Study 3
Description: Change from baseline to the last hour of the study (240-300 minutes) of EGP with a pancreatic clamp. In this study, EGP will be measured as described in Study 1 and plasma insulin and glucagon concentrations will be clamped at the basal level using the pancreatic clamp technique. Plasma glucose concentration will be allowed to decrease spontaneously after dapagliflozin or placebo administration. Somastatin will be infused with glucagon and insulin to replace basal plasma glucagon and insulin until study end.VIn this study, EGP will be measured as described in Study 1 and plasma insulin and glucagon concentrations will be clamped at the basal level using the pancreatic clamp technique. Plasma glucose concentration will be allowed to decrease spontaneously after dapagliflozin or placebo administration. Somastatin will be infused with glucagon and insulin to replace basal plasma glucagon and insulin until study end.
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: mg/kg.min
Groups:
- Dapagliflozin 10mg: Change in EGP (endogenous glucose production) after dapagliflozin administration using a pancreatic clamp
- Placebo: Change in EGP concentration after placebo administration using a pancreatic clamp
Arm/Group | Dapagliflozin 10mg | Placebo
Number analyzed (Participants) | 20 | 10
mg/kg.min | -0.23 (0.09) | -0.48 (0.05)

7. Secondary Outcome: Change in Plasma Insulin Concentrations: Study 1
Description: Plasma insulin concentrations during measurement of EGP
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: microUnits/mL
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma insulin level is measured at baseline minus the last hour of the study.
- Placebo: Subjects will receive placebo. Change in plasma insulin level is measured at baseline minus the last hour of the study.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
microUnits/mL | 5 (1) | 3 (1)

8. Secondary Outcome: Plasma Insulin Concentrations During Measurement of EGP Plus Glucose Clamp: Study 2
Description: Plasma insulin concentration is measured from baseline to the last hour of the study while using a glucose clamp. The glucose clamp technique is achieved by increase plasma glucose concentration to 125 mg/dl above basal levels by a continuous infusion of glucose. This hyperglycemic plateau is maintained by adjustment of a variable glucose infusion, based on the rate of insulin secretion and glucose metabolism. Because the plasma glucose concentration is held constant, the glucose infusion rate is an index of insulin secretion and glucose metabolism. The 3-3H-glucose infusion will be started at 6 AM to measure the basal rate of EGP. After a 3 hour tracer equilibration period (at 9 AM) subjects will receive dapagliflozin (10 mg) or placebo, and the plasma glucose conc will be measured every 5 minutes for 5 hours (from 9AM to 2 PM)
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: microUnits/mL
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma insulin level is measured at baseline minus the last hour of the study while using glucose clamp.
- Placebo: Subjects will receive placebo. Change in plasma insulin level is measured at baseline minus the last hour of the study while using glucose clamp.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
microUnits/mL | 0 (1) | 0 (1)

9. Secondary Outcome: Change in Plasma Insulin While Using Pancreatic Clamp: Study 3
Description: Plasma insulin concentration during measurement of EGP while using pancreatic clamp. In this study, EGP will be measured as described in Study 1 and plasma insulin and glucagon concentrations will be clamped at the basal level using the pancreatic clamp technique. Plasma glucose concentration will be allowed to decrease spontaneously after dapagliflozin or placebo administration. Somastatin will be infused with glucagon and insulin to replace basal plasma glucagon and insulin until study end.
Time Frame: Baseline to last hour of the study
Measure: Mean (Standard Deviation); unit: microUnits/mL
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma insulin level is measured at baseline minus the last hour of the study while using pancreatic clamp.
- Placebo: Subjects will receive placebo. Change in plasma insulin level is measured at baseline minus the last hour of the study while using pancreatic clamp.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
microUnits/mL | 2 (1) | 0 (1)

10. Secondary Outcome: Change in Glucagon: Study 1
Description: Change in glucagon concentrations during measurement of EGP
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma glucagon level is measured at baseline minus the last hour of the study.
- Placebo: Subjects will receive placebo. Change in plasma glucagon level is measured at baseline minus the last hour of the study.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
ng/ml | 5 (2) | -1 (2)

11. Secondary Outcome: Change in Glucagon Using Glucose Clamp: Study 2
Description: Plasma glucagon concentration during measurement of EGP using a glucose clamp. The glucose clamp technique is achieved by increase plasma glucose concentration to 125 mg/dl above basal levels by a continuous infusion of glucose. This hyperglycemic plateau is maintained by adjustment of a variable glucose infusion, based on the rate of insulin secretion and glucose metabolism. Because the plasma glucose concentration is held constant, the glucose infusion rate is an index of insulin secretion and glucose metabolism.
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma glucagon level is measured at baseline minus the last hour of the study while using a glucose clamp.
- Placebo: Subjects will receive placebo. Change in plasma glucagon level is measured at baseline minus the last hour of the study while using a glucose clamp.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
ng/ml | -6 (2) | -7 (3)

12. Secondary Outcome: Change in Glucagon Using Pancreatic Clamp: Study 3
Description: Measurement of change in plasma glucagon from baseline to one hour prior to end of study while using a pancreatic clamp. In this study, EGP will be measured as described in Study 1 and plasma insulin and glucagon concentrations will be clamped at the basal level using the pancreatic clamp technique. Plasma glucose concentration will be allowed to decrease spontaneously after dapagliflozin or placebo administration. Somastatin will be infused with glucagon and insulin to replace basal plasma glucagon and insulin until study end.
Time Frame: Baseline to 240-300 minutes
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Dapagliflozin: Subjects will receive dapagliflozin 10mg. Change in plasma glucagon level is measured at baseline minus the last hour of the study while using a pancreatic clamp.
- Placebo: Subjects will receive placebo. Change in plasma glucagon level is measured at baseline minus the last hour of the study while using a pancreatic clamp.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 20 | 10
ng/ml | -1 (1) | -2 (2)

ADVERSE EVENTS:
Time Frame: On each study day: Study start at 6am until study ends at 2pm.
Groups:
- Dapagliflozin: 20 subjects will receive dapagliflozin 10mg
  Dapagliflozin: Three 5-hour measurements (after dapagliflozin 10mg administration) of endogenous glucose production (EGP) will be performed on separate days.
- Placebo: 10 subjects will receive placebo
  Placebo: Three 5-hour measurements (after placebo administration) of endogenous glucose production (EGP) will be performed on separate days.
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT02984644/Prot_SAP_000.pdf